CLINICAL TRIAL: NCT04617639
Title: The Norwegian Trial of Physical Exercise After Myocardial Infarction. A Nationwide Randomized Clinical Trial After Myocardial Infarction to Determine the Effects of Supervised Physical Activity on Long-term Mortality and Morbidity
Brief Title: The Norwegian Trial of Physical Exercise After Myocardial Infarction
Acronym: NorEx
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Universitetssykehuset i Nord-Norge Hospital Trust (Unknown); Helse Bergen Hospital Trust (Unknown); Helse Sorlandet Hospital Trust (Unknown); Finnmark Hospital Trust (Other); Helgelandssykehuset Hospital Trust (Unknown); Nordlandssykehuset Hospital Trust (Unknown); Helse Fonna Hospital Trust (Unknown); Helse Forde Hospital Trust (Unknown); Helse Møre og Romsdal Hospital Trust (Unknown); Helse Nord-Trøndelag HF (Other); Akershus University Hospital Trust (Unknown); Diakonhjemmet Hospital AS (Unknown); Sykehuset Innlandet Hospital Trust (Unknown); Sykehuset Telemark Hospital Trust (Unknown); Sykehuset i Vestfold Hospital Trust (Unknown); Helse Stavanger Hospital Trust (Unknown); Vestre Viken Hospital Trust (Other); Helse Midt-Norge Hospital Trust (Unknown); University of Oslo (Other); University of Bergen (Other); University of Tromso (Other); Haraldsplass Hospital AS (Unknown); Lovisenberg Hospital AS (Unknown); Sykehuset Ostvold Hospital Trust (Unknown); St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12128; 287618 (Other Grant/Funding Number: Research Council of Norway); 287380 (Other Grant/Funding Number: Research Council of Norway)
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction
Keywords: Exercise therapy; Secondary prevention
MeSH Terms: conditions — Myocardial Infarction | interventions — Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial with blinded endpoint evaluation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical exercise (Experimental): Supervised home-based and community-based physical exercise with a dose required to increase cardiorespiratory fitness, i.e. intensity, duration and frequency that accumulates to at least 115 minutes a week of exercise, divided into at least 20 minutes a week of high/vigorous intensity physical activity (active minutes at about 85% of peak heart rate or Rated Perceived Exertion [RPE] of about 16 on Borg scale) and 95 minutes a week at moderate-intensity physical activity (active minutes at about 70% of peak heart rate or RPE of about 13 on Borg Scale), or continuous heart rate measurements amounting to at least 100 Personal Activity Intelligence (PAI) equivalents per week.
  Interventions: Behavioral: Physical exercise
- Control group I (Active Comparator): Standard care, i.e. advice at study start to follow international guidelines of moderate to vigorous physical activity intensity without further guidance and follow-up by study personnel.
  Interventions: Behavioral: Standard care
- Control group II (observation group) (Other): Follow-up through mandatory national heath registries for primary endpoint, without any contact by study personnel.
  Interventions: Behavioral: Observation group

INTERVENTIONS:
Behavioral: Physical exercise — Supervised home-based and community-based physical exercise with a dose required to increase cardiorespiratory fitness, i.e. intensity, duration and frequency that accumulates to at least 115 minutes a week of exercise, divided into at least 20 minutes a week of high/vigorous intensity physical activity (active minutes at about 85% of peak heart rate or Rated Perceived Exertion [RPE] of about 16 on Borg scale) and 95 minutes a week at moderate-intensity physical activity (active minutes at about 70% of peak heart rate or RPE of about 13 on Borg Scale), or continuous heart rate measurements amounting to at least 100 Personal Activity Intelligence (PAI) equivalents per week.
  Arms: Physical exercise
Behavioral: Standard care — Standard care, i.e. advice at study start to follow international guidelines of moderate to vigorous physical activity intensity without further guidance and follow-up by study personnel.
  Arms: Control group I
Behavioral: Observation group — Follow-up through mandatory national heath registries for primary endpoint, without any contact by study personnel
  Arms: Control group II (observation group)

SUMMARY:
Myocardial infarction (MI) remains the main cause of death in Europe with about 2 million deaths annually. According to WHO, 30 % of deaths caused by MI could be prevented if the populations adhere to official guidelines for physical activity. However, secondary prevention trials in MI patients have been of insufficient size or quality to provide conclusive evidence that physical activity reduces the risk of death or recurrent cardiovascular diseases. NorEx is the first study able to provide such evidence.

NorEx is a registry-based prospective, three-arm, randomized multicenter secondary prevention clinical trial with blinded end-point evaluation (PROBE design). The aim of the study is to investigate whether, and to what extent, moderate to high intensity supervised physical activity will reduce the risk of recurrent cardiovascular disease and death among people who have suffered a myocardial infarction. The intervention group consists of Approximately 3185 participants who will be trained to exercise for 4 years under supervision of a personal trainer. The study design includes two control groups each consisting of approximately 3200 patients.The primary composite endpoint is time to all-cause death, nonfatal acute myocardial infarction or nonfatal stroke, whatever comes first during 4 years of follow-up. The study is powered to detect a 20 % difference in the incidence of the primary endpoint between the intervention group and the control groups. Novel health IT technology was specifically designed for NorEx, including a smart watch, a NorEx mobile application and a manager portal which allows the trainers to interact with the participants. Follow-up of the participants will be through national health registries for up to 10 years after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized in a Norwegian hospital with an acute myocardial infarction (Type I) during 2013-2022. Patients are included minimum 3 months after hospitalization when they are in a stable clinical condition.
2. Norwegian national identification number
3. Able to communicate in Norwegian or other Scandinavian language
4. Being able to be physically active according to study protocol, as determined by study personnel.
5. Signed informed consent.

Exclusion criteria:

1. Persons who already participate in physical activity at a similar or higher level than what is prescribed for the intervention group, as determined by study personnel.
2. Participating or plans to participate in endurance sport competitions.
3. Expected to emigrate during the study
4. Cognitive impairment/dementia.
5. Alcohol or drug abuse, or serious psychiatric disease.
6. Known cardiac disease that may represent a contraindication for moderate or high-intensity physical activity, such as symptomatic valvular heart disease, hypertrophic cardiomyopathy, uncontrolled hypertension, in-compensated heart failure, serious arrythmia not under control after treatment, pulmonary hypertension, significant angina after revascularization and optimal drug treatment.
7. Renal insufficiency requiring dialysis.
8. Any end-stage somatic disease with short life expectancy or that is expected to interfere with the participants' ability to comply with the study protocol, such as advanced cancer, chronic lung disease with exacerbations, or other disease, as determined by study personnel.
9. Inability to comply with the study protocol due to any physical disability, somatic disease or mental problem, as determined by study personnel.
10. Residing in nursing home or other institution.
11. Participation in another trial with exercise as an intervention modality.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9700 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause mortality, or nonfatal myocardial infarction, or nonfatal stroke, whichever comes first. | 4 years
  Mortality will be assessed by linkage to the Norwegian Cause of Death Register with the use of a unique 11-digit Norwegian national identification number for each patient. The Cause of Death Register is completed by law for all deaths. Nonfatal myocardial infarction and nonfatal stroke are assessed by linkage to The Norwegian Myocardial Infarction Register and the Norwegian Stroke Register, with the use of a unique 11-digit Norwegian national identification number for each patient. All Norwegian hospitals are required by law to complete these registers for hospitalized patients.

SECONDARY OUTCOMES:
Time to all-cause mortality, or nonfatal myocardial infarction, or nonfatal stroke, whichever comes first. | 10 years
  Mortality will be assessed by linkage to the Norwegian Cause of Death Register with the use of a unique 11-digit Norwegian national identification number for each patient. The Cause of Death Register is completed by law for all deaths. Nonfatal myocardial infarction and nonfatal stroke are assessed by linkage to The Norwegian Myocardial Infarction Register and the Norwegian Stroke Register, with the use of a unique 11-digit Norwegian national identification number for each patient. All Norwegian hospitals are required by law to complete these registers for hospitalized patients.
Time to all-cause mortality, cardiac death, vascular death, noncardiovascular death, death from cancer. | 4 years and 10 years
  Mortality will be assessed by linkage to the Norwegian Cause of Death Register with the use of a unique 11-digit Norwegian national identification number for each patient. The Cause of Death Register is completed by law for all deaths.
Time to hospitalization with a diagnosis of nonfatal myocardial infarction, stroke, unstable angina pectoris, atrial fibrillation, or psychiatric disease, or a coronary revascularization procedure, or any hospitalization. | 4 years and 10 years
  Information about hospitalizations and the discharge diagnoses will be collected by means of electronic linkage to the Norwegian Patient Registry with the use of a unique 11-digit Norwegian national identification number for each patient. The Norwegian National Patient Registry includes the codes of the International Classification of Diseases, 10th Revision (ICD-10), with respect to all the main diagnoses and up to 20 secondary diagnoses and all the procedure codes from all hospitalizations in Norway.
Change in health related quality of life | Study start, 4 years and 10 years
  HeartQoL questionnaire is a core ischemic heart disease specific health related quality of life questionnaire (HRQL). The questionnaire comprises 14-items with 10-item physical and 4-item emotional subscales which are scored from 0 (poor HRQL) to 3 (better HRQL) with a global score if need.
Change in anxiety and depression | Study start, 4 and 10 years
  The Hospital Anxiety and Depression Scale (HADS) measure symptoms of anxiety and depression. The HADS is a 14 item scale where seven of the items relate to anxiety and seven relate to depression.The respondent rates each item on a 4-point scale from 0 (absence) to 3 (extreme presence). The total score is 42 (21 per subscale).
Physical and mental dimensions of health | Study start, 4 years and 10 years
  RAND-12 measures physical and mental dimensions of health. The 12 items in the questionnaire correspond to eight principal physical and mental health domains. The 12 items are summarized into two scores, a "Physical Health Summary Measure (PCS-physical component score)" and a "Mental Health Summary Measure (MCS-mental component score).
  .
Changes in insomnia | Study start, 4 years and 10 years
  The Bergen Insomnia Scale measure sleeping pattern and insomnia. The 6 items in the questionnaire are scored from 0 (absence) to 7 (every night) and are summarized to a total score with a max value between 0 (no insomnia) to 42 (extreme insomnia).
The number of consultations with a primary health care physician during the study | 4 and 10 years
  The number of consultations in primary health care will be collected by linkage to the Norwegian KUHR database with the use of a unique 11-digit Norwegian national identification number for each patient.
Use of prescription drugs | 4 and 10 years
  Use of prescription drugs during the study will be collected by linkage to the Norwegian Drug Prescription Database with the use of a unique 11-digit Norwegian national identification number for each patient.
Change in memory | 4 and 10 years
  The following 8 questions about memory will be administered by a self-administered questionnaire at start of the study and after 3.5 year and 10 years:
  1. Do you have problems with the memory?
  2. Are these problems worse than among other people on your age?
  3. Do have problems with remembering other persons name?
  4. Do have problems with following a conversation?
  5. Do have problems with remembering what happened a few minutes ago?
  6. Do have problems with doing what you have planned to do? 7 Do have problems with remembering dates?
  8. Do have problems with remembering events that took place a few days ago? The response categories for all questions are: "Never (0)", "Little or sometimes (1)", or "Often (2)".
  The scores for question 3 to 8 may be summarized to a total score between 0 (No memory problems) and 18 (severe memory problems).
Change in peak oxygen uptake (VO2peak) (mL/kg/min) | Study start, 1 year, 4 years
  Peak oxygen uptake will be measured with standard equipment for indirect calorimetry in an incremental protocol until exhaustion on either a treadmill or a bicycle ergometer. Measurements will be performed each year during the study in random samples of 150 participants in the experimental physical exercise arm and 150 participants in the active comparator arm (control group I)
Physical activity | Study start, 4 years, 10 years
  A self-administered questionnaire with questions about frequency of weekly physical activity, intensity level, and amount of weekly physical activity will be administered at baseline and end of study (3.5 years). The questionnaire consist of the following 6 questions:
  How many times do you exercise per week? (4 response categories). If you exercise 1 time or more per week, at what intensity level do you usually exercise (3 response categories).
  How many minutes do you usually exercise each time (4 response categories) How many hours per day do you spend in a sitting position ( number of hours) Do you participate in endurance sport competitions? (no, yes)

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology; Kaare Bønaa, MD prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital Clinic of Cardiology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
To be decided

REFERENCES:
- [Derived] Svenningsen A, Soderstrom S, Bucher Sandbakk S, Gullestad L, Bonaa KH, Wisloff U, Hollekim-Strand SM. Mind the intention-behavior gap: a qualitative study of post-myocardial infarction patients' beliefs and experiences with long-term supervised and self-monitored physical exercise. BMC Sports Sci Med Rehabil. 2024 Sep 27;16(1):204. doi: 10.1186/s13102-024-00987-2. PMID 39334432